CLINICAL TRIAL: NCT03028402
Title: Adjacent Segment Mechanics in Cervical Arthrodesis Patients
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, William Anderst, Associate Professor, University of Pittsburgh
Other Study IDs: STUDY19070070
Record Dates: First submitted 2016-02-10; First posted 2017-01-23 (Estimated); Last update posted 2025-02-06 (Actual); Status verified 2024-09

CONDITIONS: Intervertebral Disc Degeneration
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (5):
- Asymptomatic Controls: Individuals who have no history of neck pain, trauma or surgery, similar in age and sex to the surgical patients
- C5-C6 arthrodesis: Patients scheduled to undergo C5-C6 anterior cervical arthrodesis
  Interventions: Procedure: C5-C6 arthrodesis
- C6-C7 arthrodesis: Patients scheduled to undergo C6-C7 anterior cervical arthrodesis
  Interventions: Procedure: C5-C6 arthrodesis
- C4-C5-C6 arthrodesis: Patients scheduled to undergo C4-C5-C6 anterior cervical arthrodesis
  Interventions: Procedure: C5-C6 arthrodesis
- C5-C6-C7 arthrodesis: Patients scheduled to undergo C5-C6-C7 anterior cervical arthrodesis
  Interventions: Procedure: C5-C6 arthrodesis

INTERVENTIONS:
Procedure: C5-C6 arthrodesis — A standard Smith Robinson anterior medial approach to the cervical spine. Vertebral endplates will be prepared by removing the cartilage endplate. Tricortical anterior iliac crest autografts will be harvested with a low-speed oscillating saw. Allografts will be fresh-frozen, vacuum-sealed, nonradiated tricortical grafts. All grafts will be fashioned in a typical Smith-Robinson formation. The motion segment will be distracted approximately 2-mm beyond the graft height before the insertion of each graft. Fusion plate will be contoured to cervical lordosis. Cervical plates will be positioned using surgical midline markers. All rigid anterior plate fixations will be performed using titanium anterior fixed-angle screw systems.
  Groups: C4-C5-C6 arthrodesis; C5-C6 arthrodesis; C5-C6-C7 arthrodesis; C6-C7 arthrodesis

SUMMARY:
This study aims to determine to what extent patient-specific factors, iatrogenic factors, and biomechanical factors influence cervical spine mechanics after single-level and two-level arthrodesis.

DETAILED DESCRIPTION:
The etiology of adjacent segment pathology following cervical fusion remains highly controversial. Adjacent segment disease is believed to result from one or more of the following distinct causes:

1. the natural history of the adjacent disc;
2. disruption of the adjacent segment anatomy due to the initial surgery; and
3. biomechanical stress on the adjacent level following the fusion.

The long-term goal of our research is to reduce or prevent symptomatic adjacent segment degeneration in the spine. The overall hypothesis of this study is that adjacent segment kinematics (i.e. translations, rotations, helical axis of motion) and arthrokinematics (i.e. disc deformation and facet joint surface interactions) after ACDF are determined primarily by patient-specific anatomy and iatrogenic factors, and not by increased biomechanical stress due to the fusion.

A prospective longitudinal study is proposed to determine to what extent patient-specific factors (Specific Aim 1), iatrogenic factors (Specific Aim 2), and altered biomechanics (Specific Aim 3) affect dynamic cervical spine function following fusion. Participants will be C56 (n=22) and C67 (n=22) single-level fusion patients, C456 (n=22) and C567 (n=22) two-level fusion patients, and asymptomatic controls similar in age to the fusion patients (n=22). Patients will be tested prior to surgery, one year post-surgery, and three years post-surgery. At each test, participants will complete clinical questionnaires to assess pain and function, and they will perform full range of motion flexion\extension and axial rotation of the head and cervical spine while biplane radiographs are recorded at 30 images per second. A highly accurate and validated volumetric model-based tracking process and custom data analysis software will be utilized to determine intervertebral kinematics (i.e. translations, rotations, helical axis of motion) and arthrokinematics (i.e. disc deformation and facet joint surface interactions) at each test session.

This prospective study will identify the factors that have the greatest effect on adjacent segment mechanics after cervical fusion. If the hypotheses are confirmed, this will provide support for increased attention to patient-specific factors and surgical technique. Alternatively, if the results indicate that adjacent segment mechanics are influenced primarily by increased stress after arthrodesis, this will provide support for increased attention to the design of motion-sparing devices.

ELIGIBILITY:
Inclusion Criteria:

* Patients must agree to return for all follow-up visits and provide informed consent.
* Control subjects will be asymptomatic, with no injury or disease that will interfere with spine function, such as previous spine surgery or trauma.

Exclusion Criteria:

* Participants will have no other injury or disease that will interfere with spine function, such as previous spine surgery or trauma
* Individuals who have been previously clinically diagnosed with poor bone quality and those who do not intend to stay in the Pittsburgh area for a period of at least 3 years post-surgery will be excluded.
* Females who are pregnant or plan to be pregnant within 3 years of surgery will be excluded.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients will be between 21 and 60 years of age and will be scheduled to undergo single-level or two-level anterior cervical discectomy and fusion (ACDF) at the C56, C67, C456 or C567 levels. Indications for surgical intervention will be progressive symptoms refractory to conservative treatment for myelopathy, radiculopathy, or myeloradiculopathy resulting from degenerative spondylosis, symptomatic cervical disc herniation, or symptomatic disc degeneration.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Kinematics | pre-surgery to 3 years post-surgery
  range of motion (ROM) in degrees
Iatrogenic factors | pre-surgery to 3 years post-surgery
  adjacent segment disc height and sagittal alignment; graft height, plate placement
Kinematics | pre-surgery to 3 years post-surgery
  The helical axis of motion (HAM)
Kinematics | pre-surgery to 3 years post-surgery
  The continuous 3D intervertebral kinematics (translations and rotations).
Arthrokinematics | pre-surgery to 3 years post-surgery
  Disc deformation
Arthrokinematics | pre-surgery to 3 years post-surgery
  Facet joint capsule deformation

CONTACTS AND LOCATIONS:
Overall Officials: William Anderst, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Biodynamics Lab, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No